CLINICAL TRIAL: NCT03377712
Title: SURGICAL REPERCUSSIONS IN RESPIRATORY SYSTEM, TRUNK BIOMECHANICAL, FUNCTIONAL CAPACITY AND QUALITY OF LIFE IN PATIENTS WITH POST-TRAUMATIC BRACHIAL PLEXUS INJURIES: A PROSPECTIVE COHORT STUDY
Brief Title: Surgical Repercussions in Respiratory System in Patients With Post-Traumatic Brachial Plexus Injuries: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helen Fisio, Doctor student, Universidade Federal de Pernambuco
Other Study IDs: UFPE POSNEURO
Record Dates: First submitted 2017-12-03; First posted 2017-12-19 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Brachial Plexus Injury; Respiratory Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brachial Plexus Injury group: Patients who will be submitted to the surgical procedure and monitored for the repercussions of the surgery. Interventions: optoelectronic plethysmography, diaphragmatic ultrasound, postural evaluation, functional capacity, pain evaluation, function and quality of life
  Interventions: Device: optoelectronic plethysmography; Device: diaphragmatic ultrasound; Device: Postural evaluation; Device: Pain evaluation; Device: Evaluation of the function; Device: Functional capacity assessment; Device: Quality of life assessment
- Paired group: Healthy individuals who will be matched by sex and age with the group of patients who will effectively undergo the surgical process. Interventions: optoelectronic plethysmography, diaphragmatic ultrasound, postural evaluation and functional capacity.
  Interventions: Device: optoelectronic plethysmography; Device: diaphragmatic ultrasound; Device: Postural evaluation

INTERVENTIONS:
Device: optoelectronic plethysmography — Evaluates the thoracoabdominal kinematics and the ventilatory pattern of the patient through the filming with cameras, simple and non-invasive examinations
Device: diaphragmatic ultrasound — Evaluates the diaphragmatic mobility through images, simple and non-invasive use
Device: Postural evaluation — Evaluates the patient's posture through photos and filming, rapid examination, simple and non-invasive
Device: Pain evaluation — by means of questionnaires
  Groups: Brachial Plexus Injury group
Device: Evaluation of the function — through questionnaires
  Groups: Brachial Plexus Injury group
Device: Functional capacity assessment — Evaluated through the six-minute walk test, where the patient walks along a 30-meter corridor, simple, fast and safe assessment
  Groups: Brachial Plexus Injury group
Device: Quality of life assessment — through questionnaire
  Groups: Brachial Plexus Injury group

SUMMARY:
To evaluate the surgical repercussions in patients with traumatic brachial plexus injury in the respiratory and motor systems, trunk biomechanics, functional capacity and quality of life.

DETAILED DESCRIPTION:
Type of study will be a prospective cohort. The study will be performed at the Laboratory of Cardiopulmonary Physiotherapy of the Federal University of Pernambuco (UFPE). The sample will be calculated from a pilot study to be previously performed. The pilot study should have 10 individuals, 5 patients in each of the two groups. A group of patients who has brachial plexus injury and a group of healthy individuals for the pairing by sex and age. Eligibility criteria: patients who will undergo surgical intervention (within one year of the trauma), of both sexes, between 20 and 45 years of age, sedentary (oriented and encouraged to perform the activities of daily living at home, however , outside of any rehabilitation program) and encouraged to refrain from using tobacco. Patients with pulmonary contusions, severe pneumopathies, patients with congestive heart failure (NYHA class III or IV), diabetes mellitus, coronary artery disease, hemodynamic instability (MAP <60 mmHg), multiple thorax fractures, amputation of one limb cognitive changes. Physiotherapeutic evaluations will be performed by a single physiotherapist trained in the preoperative one, three and six months after surgery for brachial plexus injury. The instruments of evaluation included are: optoelectronic plethysmography, spirometry, manovacuometry, diaphragmatic ultrasound, g-walk, upper limb dynamometry, pain questionnaires (Mcgill and DN4), upper limb functionality questionnaire (DASH) minutes and the quality of life questionnaire (Whoquol). Expected Results: The greatest impact should be to assist the patient in the prevention and physiotherapeutic treatment in relation to the possible sequels arising from the surgical process, besides fomenting the literature, expanding the knowledge about the subject and determining the applicability of the existing therapeutic resources, so that these are not used indiscriminately in daily practice.

ELIGIBILITY:
Inclusion Criteria Patients who will undergo surgical intervention; male; between 20 and 45 years of age; sedentary.

Exclusion Criteria Pulmonary contusions; Severe pneumopathies; Diabetes mellitus; Coronary artery disease; Multiple thorax fractures; Amputation of one limb; Cognitive changes

-

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be composed of patients diagnosed with traumatic injury of the brachial plexus, at most one year of injury after the accident, confirmed by electromyography (ENMG), and who will undergo surgical intervention. The patients will be screened at the main reference center in Pernambuco, Recife Hospital / Recife
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
thoracoabdominal kinematics | There will be two evaluations: one evaluation before surgery, another after six month
  It will be evaluated through optoelectronic plethysmography
mobility diaphragmatic | There will be two evaluations: one evaluation before surgery, another after six month
  It will be evaluated by means of an ultrasound

SECONDARY OUTCOMES:
Postural evaluation | There will be two evaluations: one evaluation before surgery, another after six month
  evaluates the patient's posture through photos, rapid examination, simple and non-invasive. Only the registration of images will be reactivated
Pain | There will be two evaluations: one evaluation before surgery, another after six month
  evaluation by means of questionnaire
Evaluation of the function | There will be two evaluations: one evaluation before surgery, another after six month
  through questionnaire - Arm, Shoulder and Hand Disability (DASH). The score is given by a formula: Sum of the first 30 questions, subtract 30 and then divide by 1.2 The higher the score, the worse the function of the upper limbs (always evaluating the two limbs at the same time).
Functional capacity assessment | There will be four evaluations: one evaluation before surgery, another with one month, three and six months after the surgery
  Evaluated through the six-minute walk test, where the patient walks along a 30-meter corridor, simple, fast and safe assessment
Quality of life assessment | There will be two evaluations: one evaluation before surgery, another after six month
  through questionnaire - World Health Organization Quality of Life Instrument (WHOQOL-Brief) - DOMAINS: Physical, Psychological, Social Relations, Environment and Self-evaluation of QOL. Score the higher the score, the better the quality of life of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Helen Fuzari, Recife, Pernambuco, Brazil